CLINICAL TRIAL: NCT04204161
Title: A Clinical Study Evaluating the Safety and Efficacy of CAR-T19/CAR-T22 Treatment for Children With CD19 Positive Relapse or Refractory Childhood Acute Lymphoblastic Leukemia and Lymphoma
Brief Title: A Clinical Study of CAR-T Cells Treatment for Children With CD19+/CD22+ R/R ALL and Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen BinDeBio Ltd. (Industry)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019XY-BDB011
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Relapsed B-cell Acute Lymphoblastic Leukemia, Childhood; Refractory B-cell Acute Lymphoblastic Leukemia, Childhood; Relapsed/Refractory B-cell Lymphoma, Childhood
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T19/CAR-T22 (Experimental): CAR-T19/CAR-T22 (autologous T cells transduced with CD19 / 22 CAR-ζ/4-1BB vector) will be administered to children with R/R B cell Acute Lymphoblastic Leukemia (ALL) or Lymphoma as an IV infusion on days 0, 1 and 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: CAR-T19/CAR-T22

INTERVENTIONS:
Biological: CAR-T19/CAR-T22 — According to tumor burden and other conditions, patients will be treated with cyclophosphamide or fludarabine,then,CAR-T cells will be infused 48-72 hours later.The recommand dose is 1x10^5/kg-2.5x10^8/kg .

SUMMARY:
This is a single arm, open-label, uni-center, phase I study . In this study, Children withCD19+/CD22+ R/R B-cell acute lymphoblastic leukemia or lymphoma will be treated with CAR-T19/CAR-T22 Immunotherapy to determine the safety and efficacy of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD19+/CD22+ B cell malignancies who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled.

  1. no available curative treatment options (such as autologous or allogeneic SCT)
  2. If patients had receive immunotherapy, they should reach requirments:tumor recurrency or the number of B cells recovered.
  3. Patients with recurrence after hematopoietic stem cell transplantation need additional satisfaction: 1) no GvHD and not require immunosuppression;2) stem cell transplantation was completed for at least 4 months, and at least 6 months before the CART reinfusion;
  4. Patients must be willing to sign an informed consent.
  5. Age:≤18 years.
  6. survival>12 weeks
  7. Flow cytometry or IHC showed positive expression of CD19/ CD22 in tumor cells within two months.
  8. Routine blood test:hemoglobin>=90 g/L; platelet>=50×10^9/L.
  9. Liver function: ALT and AST≤2.5 (ULN) times the upper limits of normal (if abnormal liver function is mainly caused by tumor infiltration, it can ≤5 ULN), bilirubin <2.0 mg/dl.
  10. Renal function:BUN: 9-20mg / dl; serum creatinine<= 1.5 times upper limits of normal; endogenous creatinine clearance rate>=50 ml/min
  11. Negative serum antibody for EBV, CMV, HIV , syphilis, HBVa nd HCV.
  12. Cardiac function: stable hemodynamic and left ventricular ejection fraction (LVEF)>=55%.
  13. ECOG score ≤2。
  14. Adequate venous access for apheresis, and no other contraindications for leukapheresis

Exclusion Criteria:

1. ECOG >= 3.
2. Patients with history of T cell tumors .
3. organ failure:heart failure Ⅲ and Ⅳ;The liver reached grade C of child-turcotte .Renal failure and uremia;Respiratory failure;People with impaired consciousness.
4. Acute or chronic GVHD after allogeneic hematopoiesis. Hormone or immunosuppressant was used within 30 days.
5. steroid hormoneswere used before and after blood collection and infusion.
6. HIV infection or active hepatitis B or hepatitis C infection.
7. Uncontrolled active infection.
8. Enrolled to other clinical study in the last 4 weeks.
9. Subjects with systemic auto-immune disease or immunodeficiency.
10. Allergic to cytokines.
11. Definite neuropathic or psychotic patients, including authors of dementia or seizures, history of psychotropic substance abuse and unable to quit, or other substantial lesions that may increase central neurotoxicity.
12. Patients with malignant tumors of the central nervous system.
13. Lung, brain or intestinal tumor infiltrates.
14. The second tumor was found.
15. Allergic to cytokine antagonists.
16. Other patients that researchers considered unsuitable for inclusion.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events evaluated with NCI CTC AE, version 4.0 | 60 months
  Safety evaluation

SECONDARY OUTCOMES:
Overall remission rate | 60 months
  Overall remission rate consists of complete remission rate and partial remission rate of patients being treated with CAR-T19/CAR-T22
CAR-T cells testing | 60 months
  The level of CAR-T cells will be tested regularly by Real-time Quantitative Polymerase Chain Reaction Detecting System(qPCR) or Flow cytometry to evaluate the proliferation in vivo and long-term survival.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Zhonghua, Study Director — Shenzhen BinDeBio Tech Co.,Ltd
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No